CLINICAL TRIAL: NCT02845687
Title: Observational Study on Smoking Cessation and Cost Outcomes in the Duke Smoking Cessation Program
Brief Title: Study on Smoking Cessation and Cost Outcomes in the Duke Smoking Cessation Program
Status: Terminated | Type: Observational
Why Stopped: Per NIH request
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00073920; P50DA027840 (NIH)
Record Dates: First submitted 2016-07-05; First posted 2016-07-27 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Dependence
Keywords: nicotine addiction; cigarette smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: All participants are patients within the Quit at Duke Smoking Cessation Program. This is an observational study with no interventions.

SUMMARY:
The purpose of this study is to conduct an observational assessment of natural outcomes within the Duke Smoking Cessation Program (DSCP), "Quit at Duke." This assessment will include information regarding abstinence rates, changes in patient emotional state following treatment, and costs of operations. Primarily, this study will assess the financial sustainability and the cost-effectiveness of the program.

DETAILED DESCRIPTION:
The purpose of this study is to conduct an observational assessment of natural outcomes within the DSCP, "Quit at Duke." This is an observational study (n=3000) on patients being treated at the DSCP. No interventions are conducted, and data analyzed is collected in the course of clinical care at clinic visits to the Duke Smoking Cessation Program (DSCP). Phone calls are also conducted to determine response to medications and abstinence status up to 12 months following a quit attempt. Outcomes of variables including: demographic variables, evaluation responses, feasibility data, and abstinence rates will be analyzed using general regression models using an ANOVA-based design. Because no intervention is being conducted, there are no safety concerns related to the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Being treated at the Duke Smoking Cessation Program
* Fluent in written and spoken English.

Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit participants through Quit at Duke, also called the Duke Smoking Cessation Program (DSCP). The DSCP is a growing multi-clinic tobacco use treatment program. The initial clinic site is at Duke Cancer Center, but it is positioned to expand over the next several years to include several other clinic sites within the Duke University Health System (DUHS). There are no exclusion criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Biochemically confirmed continuous 30-day abstinence from smoking | 12 weeks post-Target Quit Day (TQD)
  Biochemically confirmed 30-day continuous abstinence. Abstinence is determined by a participant both reporting not smoking in the past 30 days AND a result of < 7 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent

SECONDARY OUTCOMES:
Biochemically confirmed 7-day point prevalence abstinence from smoking | 2 weeks post-TQD
  Biochemically confirmed 7-day continuous abstinence. Abstinence is determined by a participant both reporting not smoking in the past 7 days AND a result of < 7 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent
Biochemically confirmed 7-day point prevalence abstinence from smoking | 12 weeks post-TQD
  Biochemically confirmed 7-day continuous abstinence. Abstinence is determined by a participant both reporting not smoking in the past 7 days AND a result of < 7 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent
Self-report 7-day point prevalence abstinence from smoking | 1 day post-TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-report 7-day point prevalence abstinence from smoking | 1 week post-TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-report 7-day point prevalence abstinence from smoking | 6 month post-TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Self-report 7-day point prevalence abstinence from smoking | 12 month post-TQD
  7-day point prevalence abstinence as measured by phone-based, single-item self-report
Smoking reduction | 1 day post-TQD
  Smoking reduction as measured by cigarettes per day, as measured by phone-based self-report
Smoking reduction | 1 week post-TQD
  Smoking reduction as measured by cigarettes per day, as measured by phone-based self-report
Smoking reduction | 6 months post-TQD
  Smoking reduction as measured by cigarettes per day, as measured by phone-based self-report
Smoking reduction | 12 months post-TQD
  Smoking reduction as measured by cigarettes per day, as measured by phone-based self-report
Changes in stress | Baseline (pre-quit) to 2 and 12 weeks post-TQD
  Change in self-reported measures of stress, as measured by Perceived Stress Scale
Changes in anxiety | Baseline (pre-quit) to 2 and 12 weeks post-TQD
  Change in self-reported measures of anxiety, as measured by the GAD-7
Changes in depression | Baseline (pre-quit) to 2 and 12 weeks post-TQD
  Change in self-reported measures of depression, as measured by the PHQ-2
Changes in relapse predictors | Baseline (pre-quit) to 1 day post-TQD, 1 week post-TQD, 6 months post-TQD, and 12 months post-TQD
  Changes in self-reported measures on repeated non-standardized single-item question on stress, urges, and confidence assessed by phone
Overall cost of treatment in dollars per participant | 12 weeks post-TQD
cost of medical visits in dollars per abstinent participant | 12 weeks post-TQD
cost of medications per abstinent smoker | 12 weeks post-TQD
cost of behavioral intervention per abstinent smoker | 12 weeks post-TQD
cost of prescribed medications in dollars | 12 weeks post-TQD

OTHER OUTCOMES:
Feasibility: attendance records | up to 12 weeks post-TQD
  Feasibility as measured by attendance and completion of HIT and MIT assessed by attendance records taken by instructors at individual classes or sessions
Feasibility: website usage | up to 12 weeks post-TQD
  Feasibility as measured by website usage, as measured by electronically recorded login and site-based timer will record time accessing the site through each intervention
Feasibility: course evaluation | up to 12 weeks post-TQD
  Feasibility as measured by course evaluation
Feasibility: demographics | Baseline
  Feasibility as measured by demographics of patients at DSCP
Feasibility: Medications Used | 12 weeks post-TQD
  Feasibility as measured by medication use
Feasibility: Behavioral intervention used | 12 weeks post-TQD
  Feasibility as measured by behavioral intervention assignment
Feasibility: Attendance at DSCP appointments | 12 weeks post-TQD
  Feasibility as measured by attendance at DSCP appointments
Feasibility: Referral routes to DSCP | Baseline
  Feasibility as measured by referral routes to DSCP
Feasibility: Side effects | 1 day post-TQD
  Feasibility as measured by side effects, as measured by phone assessment
Feasibility: Side effects | 1 week post-TQD
  Feasibility as measured by side effects, as measured by phone assessment
Feasibility: Side effects | 6 months post-TQD
  Feasibility as measured by side effects, as measured by phone assessment
Feasibility: Side effects | 12 months post-TQD
  Feasibility as measured by side effects, as measured by phone assessment
Feasibility: medication adherence | 1 day post-TQD
  Feasibility as measured by medication adherence, as measured by phone assessment
Feasibility: medication adherence | 1 week post-TQD
  Feasibility as measured by medication adherence, as measured by phone assessment
Feasibility: medication adherence | 6 months post-TQD
  Feasibility as measured by medication adherence, as measured by phone assessment
Feasibility: medication adherence | 12 months post-TQD
  Feasibility as measured by medication adherence, as measured by phone assessment

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, MD, Principal Investigator — Duke University
Locations (1):
- Duke Smoking Cessation Program, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor GM, Lindson N, Farley A, Leinberger-Jabari A, Sawyer K, Te Water Naude R, Theodoulou A, King N, Burke C, Aveyard P. Smoking cessation for improving mental health. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD013522. doi: 10.1002/14651858.CD013522.pub2. PMID 33687070